CLINICAL TRIAL: NCT05468801
Title: Randomized, Triple-blind, Placebo Controlled Study to Evaluate the Efficacy of Individualized Homeopathic Remedies With High Grade of Pathological Similarity vs Conventional Standardized Pharmacological Treatment in Patients With Migraine.
Brief Title: Efficacy of Individualized Homeopathic Remedies on Migraine: a Randomized, Triple-blind, Placebo Controlled Study.
Acronym: HOMEOMIG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de Agudos Bernardino Rivadavia (Other Government)
Collaborators: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Samuel M. Arrues MD, MD Family Physician, Hospital General de Agudos Bernardino Rivadavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 136/18
Record Dates: First submitted 2022-07-10; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Migraine
Keywords: Migraine; Homeopathy; Individualized; Triple blind; Randomized; Clinical trial; headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Intervention Model Description: Randomized, Triple-blind, Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Remedy vials will be filled according randomized allocation in 2 number sets; one for the experimental group and two for the control group. Randomization information will be kept by the Study pharmaceutical responsible who will be the only person in possession of the sequence from the beginning of the study. Only the pharmaceutical responsible will have access to the randomization codes during the study and only in case of clinical emergency can break the code of an individual patient. The pharmaceutical responsible will never have any direct nor indirect contact with the study subjects. The The study statistician/s will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Homeopathic Remedy plus Standard Pharmacologic Treatment (Experimental): Each subject receives an individually selected homeopathic remedy (individualized homeopathic remedy) as an add on to the conventional standardized pharmacological treatment he/she is receiving prior and during study. Standardized pharmacological treatment will be monitored and approved at first hospital neurological visit and as a requirement needs to be unchanged within 3 months prior inclusion and throughout the study.
  Interventions: Other: Individualized Homeopathic Remedy
- Placebo plus Standard Pharmacologic Treatment (Placebo Comparator): Subjects receive an indistinguishable placebo plus the conventional standardized pharmacological treatment he/she is receiving prior and during study. Standardized pharmacological treatment will be monitored and approved at first hospital neurological visit and as a requirement needs to be unchanged within 3 months prior inclusion and throughout the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Individualized Homeopathic Remedy — An individualized homeopathic remedy selected for each subject according clinical homeopathic parameters will be administered daily in the form of oral globules as an add on to conventional treatment.
  Arms: Individualized Homeopathic Remedy plus Standard Pharmacologic Treatment
Other: Placebo — Placebo plus Standard Pharmacologic Treatment
  Arms: Placebo plus Standard Pharmacologic Treatment

SUMMARY:
Migraine, a chronic and often lifelong neurological disorder, is the second leading cause of years lived with disability worldwide. To reduce this global burden, concerted efforts are needed to implement and improve migraine health-care policies. Several observational studies showed significant improvement of different headaches types with homeopathy. The purpose of this study is the assessment of the efficacy of Individualized Homeopathic Remedies (specific remedies for each patient) versus Conventional pharmacological treatment in patients with migraine.

DETAILED DESCRIPTION:
This is a randomized, triple-blind, placebo-controlled, parallel group study in adult subjects with diagnosis of migraine with or without aura. All patients will be assessed in a screening visit at the Study Hospital Dept. of Neurology in order to confirm and certify migraine diagnosis and evaluate correctness and stability of usual acute and preventive standardized pharmacological treatment. Patients will fulfill a 30 day baseline period to monitor headache activity, migraine related symptoms, and medication usage. Subjects agreeing to participate in the study and meeting clinical-neurological eligibility criteria will then assist to a first homeopathic consultation to assess viability of homeopathic treatment and selection of the individualized homeopathic remedy. Patients who meet both neurological and homeopathic inclusion criteria will begin a three month treatment phase. An estimated of 72 patients, calculated according to the Open-Epi program ((c) 2003, 2008 Andrew G. Dean and Kevin M. Sullivan, Atlanta, GA, USA) , will be randomized according to statistics Epidat Program (4.2 version, july 2016 Panamerican Health Organization (PHO-WHO); to receive Individualized homeopathic treatment + standard pharmacological treatment OR unidentified placebo + standard pharmacological treatment. Study homeopathic remedy or placebo will be administered for a minimum period of 12 weeks with control visits every 4 weeks to assess neurological and homeopathic evolution, adherence and possible adverse events. During the study period patients will continue filling the migraine diary collecting frequency, length and type of headaches, acute medication usage and migraine associated symptoms. At the end of treatment, a final clinical homeopathic visit will take place as well as a final Neurological visit at study Hospital. Hospital visits are independent of clinical visits and performed by different study physicians.

After conclusion of treatment phase patients will have three more follow up visits for the assessment of clinical and homeopathic evolution, possible adverse events and general satisfaction with the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with certified diagnosis of migraine with or with out aura of at least one year of evolution according to the Subcommittee of Headaches Classification of the International Headache Association 3rd edition (ICHD-III)
* Patients receiving acute or preventive standardized pharmacological treatment for migraine for at least one year prior to study inclusion
* Patients do not have chronic migraine defined as Headache occurring on 15 or more days per month for more than 3 months, which has the features of migraine headache on at least 8 days per month (ICHD-III)
* Patients meeting ICHD-III criteria of probable medication overuse headache (MOH)
* Female patients in reproductive age that are correctly using a standardized contraceptive method
* Participants who are able to maintain a prospectively collected simple headache diary

Exclusion Criteria:

* Patients under standardized pharmacological treatment who have significantly (>50%) added or modified migraine preventive drugs doses within 3 months prior to study baseline
* Patients who have initiated or significantly (>50%) modified doses of any drug for any chronic treatment with any agent with proven analgesic action or psychiatric action (antidepressants, antipsychotics, mood stabilizers, etc) or neurological action (anticonvulsivants, antiparkinsonians, etc) within 3 months prior to study baseline
* Patients suffering any cause of secondary headache like trauma, metabolic or vascular disorders, non vascular intracranial lesions, abuse of alcohol or other psychoactive substances.
* Pregnant or probably pregnant patients according to date of last menstruation referred by the patient of more than 35 days in women with regular cycles or plasma beta sub-unit of human chorionic gonadotrophin in women with irregular menstrual cycles
* Patients with history of anaphylaxis, non controlled diabetes, severe disorders being neurological, cardiac, pulmonary and/or hepatic as well as psychosis or suicide ideation and/or attempts.
* Patients with other acute or chronic pain disorders, history of hemiplegic migraine or migraine with brain stem aura, history of cerebral-vascular accident, convulsions, severe coronary disease, non controlled hypertension or cognitive dysfunctions.
* Patients not meeting homeopathic clinical criteria of High Pathological Similitude defined as an homeopathic previous success probability for the selected homeopathic remedy of of 5 to 7 points in a probability scale of 1 to 7

  * NOTE: Please contact the investigator for additional information about Homeopathic criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of migraine attacks | Baseline - Month 3
  Assess the efficacy of chosen individualized homeopathic remedy in the preventive treatment of migraine, measuring the change in the number of weekly migraine attacks comparing baseline to the final month of the 3-month treatment period versus placebo.
Number of migraine days | Baseline - Month 3
  Assess the efficacy of chosen individualized homeopathic remedy in the preventive treatment of migraine, measuring the change in the number of monthly migraine days comparing baseline to the final month of the 3-month treatment period versus placebo.
Responder in frequency of migraine attacks | Baseline - Month 3
  Number of subjects achieving diminution in more than 50% of migraine attacks per month comparing baseline to the final month of the 3-month treatment period versus placebo
Responder in quantity of migraine days | Baseline - Month 3
  Number of subjects achieving diminution in more than 50% of migraine days per month comparing baseline to the final month of the 3-month treatment period versus placebo

SECONDARY OUTCOMES:
Migraine acute medication usage doses | Baseline - Month 3
  Assess the efficacy of chosen individualized homeopathic remedy in the preventive treatment of migraine, measured by the change of the required doses of standard pharmacological acute migraine drugs comparing baseline to the final month of the 3-month treatment period versus placebo.
Migraine Specific Quality of Life Questionnaire (MSQ) | Baseline - Month 3
  Assess the change in MSQ Questionnaire scores from baseline to end of treatment period versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel M Arrues, MD, Study Director — Researcher
Locations (1):
- Hospital Bernardino Rivadavia, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
After study conclusion individual participant data will be shared, specifically 1- clinical and neurological evolution previous to entering the study; 2- previous treatments; 3- bio psycho social and homeopathic relevant data pre and post treatment period to help understand homeopathic remedy action.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available 6 months after study termination, for a 12 months period.
Access Criteria: Data will be shared via e-mail.

REFERENCES:
- [Background] Tassorelli C, Diener HC, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ; International Headache Society Clinical Trials Standing Committee. Guidelines of the International Headache Society for controlled trials of preventive treatment of chronic migraine in adults. Cephalalgia. 2018 Apr;38(5):815-832. doi: 10.1177/0333102418758283. Epub 2018 Mar 4. PMID 29504482
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Background] Eisenberg DM, Kessler RC, Foster C, Norlock FE, Calkins DR, Delbanco TL. Unconventional medicine in the United States. Prevalence, costs, and patterns of use. N Engl J Med. 1993 Jan 28;328(4):246-52. doi: 10.1056/NEJM199301283280406. PMID 8418405
- [Background] Steinsbekk A, Ludtke R. Patients' assessments of the effectiveness of homeopathic care in Norway: a prospective observational multicentre outcome study. Homeopathy. 2005 Jan;94(1):10-6. doi: 10.1016/j.homp.2004.11.016. PMID 15751329
- [Background] Mathie RT, Lloyd SM, Legg LA, Clausen J, Moss S, Davidson JR, Ford I. Randomised placebo-controlled trials of individualised homeopathic treatment: systematic review and meta-analysis. Syst Rev. 2014 Dec 6;3:142. doi: 10.1186/2046-4053-3-142. PMID 25480654
- [Background] Mathie RT. Controlled clinical studies of homeopathy. Homeopathy. 2015 Oct;104(4):328-32. doi: 10.1016/j.homp.2015.05.003. PMID 26678738
- [Background] Kristoffersen ES, Aaseth K, Grande RB, Lundqvist C, Russell MB. Self-reported efficacy of complementary and alternative medicine: the Akershus study of chronic headache. J Headache Pain. 2013 Apr 18;14(1):36. doi: 10.1186/1129-2377-14-36. PMID 23596996
- [Background] Danno K, Colas A, Masson JL, Bordet MF. Homeopathic treatment of migraine in children: results of a prospective, multicenter, observational study. J Altern Complement Med. 2013 Feb;19(2):119-23. doi: 10.1089/acm.2011.0821. Epub 2012 Sep 14. PMID 22978244
- [Background] Owen JM, Green BN. Homeopathic treatment of headaches: a systematic review of the literature. J Chiropr Med. 2004 Spring;3(2):45-52. doi: 10.1016/S0899-3467(07)60085-8. PMID 19674623
- [Background] Mathie RT, Roniger H, Van Wassenhoven M, Frye J, Jacobs J, Oberbaum M, Bordet MF, Nayak C, Chaufferin G, Ives JA, Dantas F, Fisher P. Method for appraising model validity of randomised controlled trials of homeopathic treatment: multi-rater concordance study. BMC Med Res Methodol. 2012 Apr 17;12:49. doi: 10.1186/1471-2288-12-49. PMID 22510227
- [Background] Bell IR, Lewis DA 2nd, Brooks AJ, Schwartz GE, Lewis SE, Walsh BT, Baldwin CM. Improved clinical status in fibromyalgia patients treated with individualized homeopathic remedies versus placebo. Rheumatology (Oxford). 2004 May;43(5):577-82. doi: 10.1093/rheumatology/keh111. Epub 2004 Jan 20. PMID 14734789
- [Background] Aghadiuno M. A study of the inter-observer reliability of paper case analysis. Homeopathy. 2002 Jan;91(1):10-7. doi: 10.1054/homp.2001.0016. PMID 12371444
- [Background] Brien S, Prescott P, Owen D, Lewith G. How do homeopaths make decisions? An exploratory study of inter-rater reliability and intuition in the decision making process. Homeopathy. 2004 Jul;93(3):125-31. doi: 10.1016/j.homp.2004.04.001. PMID 15287431
- [Background] Souter K. Heuristics and bias in homeopathy. Homeopathy. 2006 Oct;95(4):237-44. doi: 10.1016/j.homp.2006.07.008. PMID 17015195
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Hepp Z, Bloudek LM, Varon SF. Systematic review of migraine prophylaxis adherence and persistence. J Manag Care Pharm. 2014 Jan;20(1):22-33. doi: 10.18553/jmcp.2014.20.1.22. PMID 24372457
- [Background] Stub T, Musial F, Kristoffersen AA, Alraek T, Liu J. Adverse effects of homeopathy, what do we know? A systematic review and meta-analysis of randomized controlled trials. Complement Ther Med. 2016 Jun;26:146-63. doi: 10.1016/j.ctim.2016.03.013. Epub 2016 Mar 26. PMID 27261996
- [Background] Ashina M, Katsarava Z, Do TP, Buse DC, Pozo-Rosich P, Ozge A, Krymchantowski AV, Lebedeva ER, Ravishankar K, Yu S, Sacco S, Ashina S, Younis S, Steiner TJ, Lipton RB. Migraine: epidemiology and systems of care. Lancet. 2021 Apr 17;397(10283):1485-1495. doi: 10.1016/S0140-6736(20)32160-7. Epub 2021 Mar 25. PMID 33773613